CLINICAL TRIAL: NCT04878055
Title: A Phase 3, Double-blind, Randomized, Placebo-controlled, Multicenter Study on the Efficacy and Safety of Reparixin in the Treatment of Hospitalized Patients With Severe COVID-19 Pneumonia
Brief Title: Study on Efficacy and Safety of Reparixin in the Treatment of Hospitalized Patients With Severe COVID-19 Pneumonia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REP0220; 2020-005919-51 (EudraCT Number)
Record Dates: First submitted 2021-04-30; First posted 2021-05-07 (Actual); Results first posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-05

CONDITIONS: Pneumonia, Viral
Keywords: Covid-19; SARS-CoV-2; Pneumonia; Severe pneumonia
MeSH Terms: conditions — Pneumonia, Viral; COVID-19; Pneumonia | interventions — reparixin

STUDY DESIGN:
Intervention Model Description: subjects will be randomized with a 2:1 randomization ratio
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reparixin (Experimental): Reparixin oral tablets, 1200 mg three times daily (TID) (2 tablets 600 mg each, TID) for up to 21 days or until decision of discharge from the hospital, on top of standard supportive care
  Interventions: Drug: Reparixin
- Placebo (Placebo Comparator): placebo, 2 tablets TID (identical to Reparixin tablets) for up to 21 days or until decision of discharge from the hospital, on top of standard supportive care.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Reparixin — 2 tablets of Reparixin (600 mg each), for the total of three daily administrations (6 tablets daily).
  Other Names: DF 1681Y
  Arms: Reparixin
Other: Placebo — Matched placebo, i.e. 2 tablets for the total of three daily administrations (6 tablets daily).
  Arms: Placebo

SUMMARY:
The study objective is to assess Efficacy and safety of Reparixin treatment as compared to placebo (both on top of standard treatment) in adult patients with severe COVID-19 pneumonia.

DETAILED DESCRIPTION:
This is a phase 3 clinical trial designed as a randomized, double-blind, placebo-controlled, multicentre study to evaluate the efficacy and safety of Reparixin in hospitalized adult patients with severe COVID-19 pneumonia.

Patients will be screened for the participation in the study and eventually randomized based on an unbalanced randomization scheme (2:1) to Reparixin oral tablets (2 x 600 mg TID) for up to 21 days or to placebo.

An unequal randomization is justified by the need to gain experience and more safety data with the investigated treatment and by an expected better acceptability of the trial by patients.

The placebo control arm is justified by the unavailability of a well-defined standard of care for subjects with COVID-19 pneumonia who are candidates for this study.

All patient will receive the standard supportive care based on the patient's clinical need. Follow-up information on the patient's clinical condition will be collected until day 90.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 90, male and female subject of any race
2. Reverse transcriptase Polymerase Chain Reaction (rt-PCR)-confirmed COVID-19 infection based on a nasal / oropharyngeal swab within 10 days before randomization
3. At least one of the following: 1) Respiratory distress with tachypnea (RR ≥ 24 breaths/min without oxygen); 2) Partial arterial oxygen pressure (PaO2) / Fraction of inspiration O2 (FiO2), P/F >100 and <300 mmHg (1mmHg = 0.133kPa), 3) SpO2 ≤ 94% while breathing ambient air.

   Calculation through validated Sat/FiO2 scales is allowed. P/F value of reference if the last available before the signature of consent.
4. Need of supplemental oxygen (i.e. new use of supplemental oxygen, or increased oxygen requirement if on chronic oxygen) requiring low- or high-flow oxygen or non-invasive mechanical ventilation (7-point WHO-OS category 4 or 5).
5. Radiological chest imaging (X-rays, CT scan) confirms lung involvement and inflammation.

Exclusion Criteria:

1. Cannot obtain informed consent.
2. Hepatic dysfunction with Child Pugh score B or C, or ALT or AST> 5 times the upper limit.
3. Renal dysfunction with estimated glomerular filtration rate (MDRD) < 50 mL/min/1.73 m2 or patient receiving continuous renal replacement therapy, hemodialysis, or peritoneal dialysis.
4. Bacterial sepsis (besides COVID-19 sepsis).
5. Known congenital or acquired immune deficiency.
6. Positive or missing pregnancy test before first drug intake or day 1; pregnant or lactating women; women of childbearing potential and fertile men who do not agree to use at least one primary form of contraception for the duration of the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2021-02-14 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Landoni, MD, PhD, Principal Investigator — Ospedale San Raffaele
Locations (17):
- United States (2):
  - The George Washington University Medical Faculty Associates, 2150 Pennsylvania Avenue NW, Washington D.C., District of Columbia
  - Franciscan Alliance, 421 N Emerson Ave,, Greenwood, Indiana
- Italy (15):
  - Policlinico S. Orsola Malpighi UO di Pneumologia e Terapia Int. Respiratoria, Bologna
  - Ospedale Policlinico San Martino Malattie infettive e tropicali, Genova
  - Ospedale regionale San Salvatore U.O.C. Anestesia e Rianimazione, L’Aquila
  - IRCCS Ospedale San Raffaele Centro di Ricerca Anestesia e Rianimazione, Milan
  - ASST SANTI PAOLO E CARLO Ospedale San Paolo Struttura Complessa Malattie Infettive, Milan
  - IRCCS Istituto Clinico Humanitas U.O. Medicina D'Urgenza, Milan
  - ASST Grande Ospedale Metropolitano Niguarda Dipartimento Malattie Infettive, Milan
  - ASST-Monza Ospedale San Gerardo Malattie Infettive, Monza
  - A.O.U. Federico II Malattie Infettive del Policlinico Federico II, Napoli
  - Università della Campania "Luigi Vanvitelli" Dipartimento di Malattie Infettive, Napoli
  - Policlinico Universitario Campus Bio-Medico UOC Anestesia e Rianimazione, Roma
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I, UOC Malattie Infettive, Roma
  - Università Cattolica del Sacro Cuore - Policlinico Universitario "Agostino Gemelli" - Istituto di Clinica delle Malattie Infettive, Roma
  - ASST dei Sette Laghi Ospedale di Circolo e Fondazione Macchi Struttura Complessa Malattie infettive e tropicali, Varese
  - A.O.U. Integrata di Verona U.O. Medicina Respiratoria, sezione di Medicina Interna, Verona

REFERENCES:
- [Derived] Piemonti L, Landoni G, Voza A, Puoti M, Gentile I, Coppola N, Nava S, Mattei A, Marinangeli F, Marchetti G, Bonfanti P, Mastroianni CM, Bassetti M, Crisafulli E, Grossi PA, Zangrillo A, Desai A, Merli M, Foggia M, Carpano M, Schiavoni L, D'Arminio Monforte A, Bisi L, Russo G, Busti F, Rovelli C, Perrotta E, Goisis G, Gavioli EM, Toya S, De Pizzol M, Mantelli F, Allegretti M, Minnella EM. Efficacy and Safety of Reparixin in Patients with Severe COVID-19 Pneumonia: A Phase 3, Randomized, Double-Blind Placebo-Controlled Study. Infect Dis Ther. 2023 Oct;12(10):2437-2456. doi: 10.1007/s40121-023-00871-5. Epub 2023 Oct 5. PMID 37798468

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The eligible patient population consisted of hospitalized adult patients with reverse transcriptase polymerase chain reaction (rt-PCR)-confirmed severe COVID-19. Patients were considered to have severe disease in the presence of respiratory distress and requiring supplemental oxygen. No gender and/or ethnicity restrictions applied.
Pre-assignment Details: A total of 287 patients were enrolled and 279 of them were randomized to the assigned treatment group (8 patients were not randomized): 185 patients were randomized to receive Reparixin and 94 patients were randomized to receive placebo (N=279). Nine of these latter were randomized but not treated (3 Reparixin and 6 Placebo). Hence, the number of treated patients (starters) was 270 (182 in Reparixin and 88 in placebo).
Groups:
- Reparixin: Reparixin oral tablets, 1200 mg three times daily (TID) (2 tablets 600 mg each, TID) for up to 21 days or until decision of discharge from the hospital, on top of standard supportive care
  Reparixin: 2 tablets of Reparixin (600 mg each), for the total of three daily administrations (6 tablets daily).
  Please note that patients randomized to Reparixin were 185, but the ones receiving at least one dose of IMP were 182. Three patients, hence, in this group were excluded from the primary FAS analysis of efficacy and from the safety analysis.
- Placebo: Placebo, 2 tablets TID (identical to Reparixin tablets) for up to 21 days or until decision of discharge from the hospital, on top of standard supportive care.
  For each administration, two tablets of Reparixin (600 mg each) or placebo were taken, for the total of three daily administrations (6 tablets daily). It was advisable to take the tablets with a glass of water to facilitate swallowing.
  Please note that patients randomized to placebo were 94, but the ones receiving it were 88. Six patients in this group, hence, were excluded from the primary FAS analysis of efficacy and from the safety analysis.
Period: Overall Study
Arm/Group | Reparixin | Placebo
Started | 182 | 88
FAS Population | 182 | 88
Completed | 147 | 70
Not Completed | 35 | 18
Not completed — Patient transferred in another department | 0 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Day 60 visit not performed by mistake | 0 | 4
Not completed — Adverse Event | 12 | 7
Not completed — Other | 5 | 0
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Lost to Follow-up | 10 | 1

BASELINE CHARACTERISTICS:
Population: FAS Full Analysis Set: set which consisted of all randomized subjects who received at least one dose of the IMP. The FAS population was analyzed according to the intent-to-treat (ITT) principle, i.e. by treatment allocation regardless the occurrence of intercurrent events (treatment policy strategy).
Groups:
- Total: Total of all reporting groups
Arm/Group | Reparixin | Placebo | Total
Number analyzed (Participants) | 182 | 88 | 270
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 112 | 58 | 170
  >=65 years | 70 | 30 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (11.8) | 60.0 (12.0) | 60.9 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 25 | 75
  Male | 132 | 63 | 195
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 22 | 72
  Not Hispanic or Latino | 132 | 66 | 198
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 182 | 88 | 270

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Alive and Free of Respiratory Failure at Day 28
Description: The event variable is defined as "the proportion of patients alive and free of respiratory failure at Day 28". This means no need of invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) or admission to intensive care unit (ICU) linked to worsening of respiratory parameters compared to baseline.
Time Frame: At day 28
Population: The Full Analysis Set (FAS), which consisted of all randomized subjects who received at least one dose of the IMP.
Measure: Number; unit: participants
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 182 | 88
participants | 152 | 71
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Analysis is based on logistic regression model with Multiple Imputation under missing not at random using retrieve dropouts with proportion of patients alive and free of respiratory failure at Day 28 as dependent variable, treatment, age group, gender and presence of concomitant disease at baseline as qualitative independent variables. Site is considered as random effects that vary randomly among patients; Test type: Superiority; p = 0.216, Two-sided regression, Logistic; Odds Ratio (OR) = 1.626, 95% CI 2-sided [0.752 to 3.514]

2. Secondary Outcome: Proportion of Patients Alive and Free of Respiratory Failure at Day 60
Description: This key secondary efficacy endpoint of the study is defined as "the proportion of patients alive and free of respiratory failure at Day 60", i.e. with no need of invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) or admission to intensive care unit (ICU) linked to worsening of respiratory parameters compared to baseline.
Time Frame: At day 60
Population: FAS population is used in this table. Discrepancies between the total number of patients in the FAS and patients actually analyzed in the logistic regression model are due to the presence of missing data for which no imputation methods are expected for this endpoint.
Measure: Number; unit: participants
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 159 | 78
participants | 141 | 66
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.377, Chi-squared; Comparison between treatment arms is performed by means of a Chi-squared test

3. Secondary Outcome: Mortality Rates up to Day 28
Description: This key secondary efficacy endpoint describes number and proportion along with the 95% CI (Clopper-Pearson's formula) of patients who died up to Day 28.
Time Frame: Up to Day 28
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 168 | 81
participants | 10 | 7
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority — Analysis is based on logistic regression model with proportion of patients died up to Date 28 as dependent variable, treatment, age group, gender and presence of concomitant disease at baseline as qualitative independent variables. Site is considered as random effects that vary randomly among patients; p = 0.17, Two-sided regression, Logistic; Odds Ratio (OR) = 0.468, 95% CI 2-sided [0.158 to 1.386]

4. Secondary Outcome: Incidence of ICU Admission Until Day 28
Description: This is a key secondary efficacy endpoint. Admissions to Intensive Care Unit (ICU) had to be considered only in presence of significant worsening of respiratory status. This condition was objectively identified by means of a decrease of PaO2/FiO2 ratio of at least 40% from the baseline value or by a worsening of Investigator's Interpretation.
Time Frame: Until day 28
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 171 | 83
participants | 27 | 18
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.168, Regression, Logistic; Odds Ratio (OR) = 0.561, 95% CI 2-sided [0.247 to 1.277]

5. Secondary Outcome: Time to Recovery (Category 1 - 2 - 3 of the 7-point WHO Ordinal Scale of Clinical Improvement (WHO-OS)) Until Day 28
Description: This is a key secondary efficacy endpoint. The event "recovery" was considered as such, if the patient has scored category 1, 2 or 3 from the 7-point WHO Ordinal Scale of clinical improvement (WHO-OS), otherwise it will be considered free of event.
  Category 1: not hospitalized, with resumption of normal activities; 2: not hospitalized, but unable to resume normal activities; 3: hospitalized, not requiring supplemental oxygen; [4: hospitalized, requiring supplemental oxygen; 5: hospitalized, requiring high-flow oxygen therapy, non-invasive mechanical ventilation, or both; 6: hospitalized, requiring ECMO, invasive mechanical ventilation, or both; 7: death]. The lower the category, the better the outcome.
Time Frame: Until Day 28
Population: The Full Analysis Set (FAS), which consisted of all randomized subjects who received at least one dose of the IMP.
Measure: Number; unit: number of patients with event (recovery)
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 182 | 88
number of patients with event (recovery) | 141 | 63
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Until Day 28; Test type: Superiority — Estimates are calculated using a nonparametric method for cumulative incidence function with competing risks data. Estimates were calculated taking into account the following competing risks: Death, discontinuation for AEs and patient transferred to another institution; p = 0.167, Gray's Test

6. Secondary Outcome: Proportion of Patients Alive and Free of Respiratory Failure at Fixed Timepoints
Description: The event variable is defined as the proportion of patients alive and free of respiratory failure at fixed timepoints. This means no need of invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) or admission to intensive care unit (ICU) linked to worsening of respiratory parameters compared to baseline.
  Admissions to ICU had to be considered only in presence of significant worsening of respiratory status.
  This condition was objectively identified by means of a decrease of PaO2/FiO2 ratio of at least 40% from the baseline value or by a worsening of Investigator's Interpretation.
Time Frame: At Days 3, 7(±1),14(±2), 21(±2) and 90(±2) after randomization (randomization = day 1)
Population: The Full Analysis Set (FAS), which consisted of all randomized subjects who received at least one dose of the IMP.
Measure: Number; unit: participants
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 182 | 88
participants
  Day 3: number analyzed (Participants) | 180 | 88
  Day 3 | 179 | 87
  Day 7 (+/-1): number analyzed (Participants) | 179 | 87
  Day 7 (+/-1) | 171 | 79
  Day 14 (+/-2): number analyzed (Participants) | 173 | 83
  Day 14 (+/-2) | 160 | 73
  Day 21 (+/-2): number analyzed (Participants) | 172 | 83
  Day 21 (+/-2) | 155 | 71
  Day 90: number analyzed (Participants) | 33 | 17
  Day 90 | 15 | 5
Statistical Analysis 1: Comparison: Reparixin vs Placebo; At Day 3 - please note that the number of subjects is 268 (180+88) and not 270; Test type: Superiority; p = 0.55, Fisher Exact — Comparison between treatment arms is performed by means of a Fisher's Exact test
Statistical Analysis 2: Comparison: Reparixin vs Placebo; At Day 7 - Please note that the total of subjects in this analysis is not 270 but 266 (n=179 in the Reparixin group and n=87 in the placebo group); Test type: Superiority; p = 0.128, Chi-squared; Comparison between treatment arms is performed by means of a Chi-squared mean
Statistical Analysis 3: Comparison: Reparixin vs Placebo; At Day 14 - Please note that the total of subjects in this analysis is not 270 but 256 (n=173 in the Reparixin group and n=83 in the placebo group); Test type: Superiority; p = 0.235, Chi-squared; Comparison between treatment arms is performed by means of a Chi-squared test
Statistical Analysis 4: Comparison: Reparixin vs Placebo; At Day 21 - Please note that the total of subjects in this analysis is not 270 but 255 (n=172 in the Reparixin group and n=83 in the placebo group); Test type: Superiority; p = 0.281, Chi-squared; Comparison between treatment arms is performed by means of a Chi-squared test
Statistical Analysis 5: Comparison: Reparixin vs Placebo; At Day 90 - Please note that the total of subjects in this analysis is not 270 but 50 (n=33 in the Reparixin group and n=17 in the placebo group); Test type: Superiority; p = 0.273, Chi-squared; Comparison between treatment arms is performed by means of a Chi-squared test

7. Secondary Outcome: Mean Changes From Baseline in Clinical Severity Score Based on the 7-point WHO-OS at Fixed Timepoints
Description: Changes from baseline in clinical severity score are analyzed based on the 7-point WHO-OS. The 7-point WHO Ordinal Scale of clinical improvement (WHO-OS), comprises the following categories: 1: not hospitalized, with resumption of normal activities; 2: not hospitalized, but unable to resume normal activities; 3: hospitalized, not requiring supplemental oxygen; 4: hospitalized, requiring supplemental oxygen; 5: hospitalized, requiring high-flow oxygen therapy, non-invasive mechanical ventilation, or both; 6: hospitalized, requiring ECMO, invasive mechanical ventilation, or both; 7: death.
Time Frame: At days 3, 7, 14, 21, 28 and End of Treatment (EoT, up to 30 days); days 60 and 90; at hospital discharge (HD, up to 2 months), and at the EoS (up to 3 months)
Population: The Full Analysis Set (FAS) consisted of all randomized subjects who received at least one dose of the IMP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 182 | 88
score on a scale
  Day 3: number analyzed (Participants) | 171 | 84
  Day 3 | -0.1 (0.4) | 0.0 (0.5)
  Day 7: number analyzed (Participants) | 166 | 80
  Day 7 | -0.4 (1.0) | -0.3 (0.9)
  Day 14: number analyzed (Participants) | 142 | 67
  Day 14 | -1.7 (1.5) | -1.5 (1.6)
  Day 21: number analyzed (Participants) | 121 | 55
  Day 21 | -2.4 (1.5) | -2.3 (1.6)
  EoT: number analyzed (Participants) | 164 | 77
  EoT | -0.9 (1.0) | -0.7 (1.1)
  Day 28: number analyzed (Participants) | 131 | 59
  Day 28 | -2.8 (1.4) | -2.6 (1.5)
  Hospital Discharge: number analyzed (Participants) | 134 | 61
  Hospital Discharge | -1.6 (0.9) | -1.6 (0.8)
  Day 60: number analyzed (Participants) | 136 | 65
  Day 60 | -3.4 (0.6) | -3.2 (0.9)
  Day 90: number analyzed (Participants) | 14 | 4
  Day 90 | -3.4 (0.6) | -3.5 (0.6)
  EOS: number analyzed (Participants) | 154 | 75
  EOS | -3.0 (1.5) | -2.6 (1.8)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; At Day 3 - Please note that the number of subjects in this analysis is not 270 but 255; Test type: Superiority; p = 0.047, Wilcoxon (Mann-Whitney) — Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test
Statistical Analysis 2: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.262, Wilcoxon (Mann-Whitney); Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test
Statistical Analysis 3: Comparison: Reparixin vs Placebo; At Day 14 - Please note that the number of subjects in this analysis is not 270 but 209; Test type: Superiority; p = 0.367, Wilcoxon (Mann-Whitney); Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test
Statistical Analysis 4: Comparison: Reparixin vs Placebo; At Day 21 - Please note that the number of subjects in this analysis is not 270 but 176; Test type: Superiority; p = 0.882, Wilcoxon (Mann-Whitney) — Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test
Statistical Analysis 5: Comparison: Reparixin vs Placebo; At Day 28 - Please note that the number of subjects in this analysis is not 270 but 190; Test type: Superiority; p = 0.19, Wilcoxon (Mann-Whitney); Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test
Statistical Analysis 6: Comparison: Reparixin vs Placebo; At Day 60 - Please note that the number of subjects in this analysis is not 270 but 201; Test type: Superiority; p = 0.161, Mann-Whitney U test — Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test
Statistical Analysis 7: Comparison: Reparixin vs Placebo; At Day 90 - Please note that the number of subjects in this analysis is not 270 but 18; Test type: Superiority; p = 0.853, Mann-Whitney U test; Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test
Statistical Analysis 8: Comparison: Reparixin vs Placebo; At EOS - Please note that the number of subjects in this analysis is not 270 but 229; Test type: Superiority; p = 0.068, Wilcoxon (Mann-Whitney); Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test
Statistical Analysis 9: Comparison: Reparixin vs Placebo; At hospital discharge (HD) - Please note that the number of subjects in this analysis is not 270 but 195; Test type: Superiority; p = 0.672, Wilcoxon (Mann-Whitney); Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test
Statistical Analysis 10: Comparison: Reparixin vs Placebo; At end of treatment (EoT) - Please note that the number of subjects in this analysis is not 270 but 241; Test type: Superiority; p = 0.153, Wilcoxon (Mann-Whitney); Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test

8. Secondary Outcome: Number of Patients With Clinical Improvement 1 up to Day 28 (Decline of 1 Category in the 7-point WHO-OS)
Description: Clinical improvement 1 is defined as the decline of 1 category in the 7-point WHO-OS up to Date 28. The clinical improvement 1 up to Day 28 was analyzed as described for time to recovery: an event was considered as such, if patient declined of at least 1 category in the 7-point WHO-OS respect to the baseline, otherwise it was be considered free of event.
Time Frame: Day 1 (baseline), Days 3, 7, 14, 21, 28.
Population: The Full Analysis Set (FAS) consisted of all randomized subjects who received at least one dose of the IMP.
Measure: Number; unit: number of patients with event
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 182 | 88
number of patients with event
  Day 1 | 0 | 0
  Day 3 | 19 | 6
  Day 7 | 56 | 22
  Day 14 | 123 | 50
  Day 21 | 146 | 66
  Day 28 | 152 | 68
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority — Estimates are calculated using a nonparametric method for cumulative incidence function with competing risks data. The null hypothesis is that the cumulative incidence functions are identical across treatment groups and estimates are calculated taking into consideration the following competing risks: Death, reasons for discontinuation for Adverse events and patient transferred to another institution; p = 0.07, Grey's test

9. Secondary Outcome: Percentage of Participants With Clinical Improvement 1 up to Day 28
Description: Clinical improvement 1 up to Date 28 for this outcome is expressed as cumulative incidence function (CIF in %). CIF allows for estimation of the occurrence of an event while taking into account the following competing risks: death, reasons for discontinuation for Adverse events and patient transferred to another institution. Estimates are calculated using a nonparametric method. The null hypothesis is that the cumulative incidence functions are identical across treatment groups.
Time Frame: At day 28
Population: The Full Analysis Set (FAS), which consisted of all randomized subjects who received at least one dose of the IMP.
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 182 | 88
% of participants | 87.2 [81.2 to 91.4] | 81.1 [70.6 to 88.2]
Statistical Analysis 1: Comparison: Reparixin vs Placebo; number of patients included in the analysis=25; Test type: Superiority; p = 0.07, Gray's test

10. Secondary Outcome: Number of Patients With Clinical Improvement 2 up to Day 28 (Decline of 2 Categories in the 7-point WHO-OS)
Description: Clinical improvement 2 is defined as the decline of 2 categories in the 7-point WHO-OS) up to Date 28. Clinical improvement 2 up to Date 28 was analyzed as described for time to recovery. An event was considered as such, if patient declined of at least 2 categories in the 7-point WHO-OS respect to the baseline, otherwise it was considered free of event.
Time Frame: Day 1 (baseline), Days 3, 7, 14, 21, 28
Population: The Full Analysis Set (FAS) consisted of all randomized subjects who received at least one dose of the IMP.
Measure: Number; unit: number of patients with event
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 182 | 88
number of patients with event
  Day 1 | 0 | 0
  Day 3 | 0 | 0
  Day 7 | 19 | 6
  Day 14 | 78 | 35
  Day 21 | 105 | 50
  Day 28 | 120 | 56
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Comparison at day 28; Test type: Superiority — Estimates are calculated using a nonparametric method for cumulative incidence function with competing risks data. The null hypothesis is that the cumulative incidence functions are identical across treatment groups and estimates are calculated taking into consideration the following competing risks: Reasons for discontinuation for Adverse events and patient transferred to another institution; p = 0.668, Gray's test

11. Secondary Outcome: Percentage of Participants With Clinical Improvement 2 up to Day 28
Description: Clinical improvement 2 up to Day 28 is defined as cumulative incidence function (CIF, in %). CIF allows for estimation of the occurrence of an event while taking into account the following competing risks: death, reasons for discontinuation for Adverse events and patient transferred to another institution. Estimates are calculated using a nonparametric method. The null hypothesis is that the cumulative incidence functions are identical across treatment groups.
Time Frame: At Day 28
Population: FAS Full Analysis Set: set which consisted of all randomized subjects who received at least one dose of the IMP. But FAS patients with at least one major (i.e. error in IMP administration, I/E criteria violation) or minor protocol deviation (i.e. not respecting visit schedule) up to Day 28 couldn't be considered in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 182 | 88
Percentage of patients | 69.9 [62.3 to 76.2] | 67.7 [56.3 to 76.7]
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Number of patients included in the analysis = 59; Test type: Superiority; p = 0.668, Gray's test

12. Secondary Outcome: Time to Discharge From Hospital up to Day 28
Description: Time to discharge from hospital up to Day 28 is analyzed as described for time to recovery.
Time Frame: Day 1 (baseline), Days 3, 7, 14, 21, 28
Population: FAS Full Analysis Set: set which consisted of all randomized subjects who received at least one dose of the IMP.
Measure: Number; unit: number of patients with event
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 182 | 88
number of patients with event
  Day 1 | 0 | 0
  Day 3 | 2 | 0
  Day 7 | 19 | 10
  Day 14 | 100 | 40
  Day 21 | 127 | 58
  Day 28 | 143 | 64
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Estimates are calculated using a nonparametric method for cumulative incidence function with competing risks data. The null hypothesis is that the cumulative incidence functions are identical across treatment groups and estimates are calculated taking into consideration the following competing risks: Reasons for discontinuation for Adverse events and patient transferred to another institution; Test type: Superiority; p = 0.23, Gray's test

13. Secondary Outcome: Clinical Status Either in Hospital or at Home (7-point WHO-OS) at Fixed Time Points
Description: Clinical status is analyzed based on the 7-point WHO-OS. The 7-point WHO Ordinal Scale of clinical improvement (WHO-OS), comprises the following categories: 1: not hospitalized, with resumption of normal activities; 2: not hospitalized, but unable to resume normal activities; 3: hospitalized, not requiring supplemental oxygen; 4: hospitalized, requiring supplemental oxygen; 5: hospitalized, requiring high-flow oxygen therapy, non-invasive mechanical ventilation, or both; 6: hospitalized, requiring ECMO, invasive mechanical ventilation, or both; 7: death. The higher the score, the worse the outcome.
Time Frame: as for outcome 7
Population: FAS Full Analysis Set: set which consisted of all randomized subjects who received at least one dose of the IMP.
Measure: Number; unit: number of patients with event
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 182 | 88
number of patients with event
  day 3 score 1: number analyzed (Participants) | 171 | 84
  day 3 score 1 | 0 | 0
  day 3 score 2: number analyzed (Participants) | 171 | 84
  day 3 score 2 | 0 | 0
  day 3 score 3: number analyzed (Participants) | 171 | 84
  day 3 score 3 | 5 | 1
  day 3 score 4: number analyzed (Participants) | 171 | 84
  day 3 score 4 | 85 | 40
  day 3 score 5: number analyzed (Participants) | 171 | 84
  day 3 score 5 | 81 | 42
  day 3 score 6: number analyzed (Participants) | 171 | 84
  day 3 score 6 | 0 | 0
  day 3 score 7: number analyzed (Participants) | 171 | 84
  day 3 score 7 | 0 | 1
  day 7 score 1: number analyzed (Participants) | 166 | 80
  day 7 score 1 | 7 | 2
  day 7 score 2: number analyzed (Participants) | 166 | 80
  day 7 score 2 | 1 | 0
  day 7 score 3: number analyzed (Participants) | 166 | 80
  day 7 score 3 | 31 | 16
  day 7 score 4: number analyzed (Participants) | 166 | 80
  day 7 score 4 | 66 | 27
  day 7 score 5: number analyzed (Participants) | 166 | 80
  day 7 score 5 | 54 | 30
  day 7 score 6: number analyzed (Participants) | 166 | 80
  day 7 score 6 | 6 | 5
  day 7 score 7: number analyzed (Participants) | 166 | 80
  day 7 score 7 | 1 | 0
  day 14 score 1: number analyzed (Participants) | 142 | 67
  day 14 score 1 | 52 | 24
  day 14 score 2: number analyzed (Participants) | 142 | 67
  day 14 score 2 | 10 | 3
  day 14 score 3: number analyzed (Participants) | 142 | 67
  day 14 score 3 | 28 | 12
  day 14 score 4: number analyzed (Participants) | 142 | 67
  day 14 score 4 | 29 | 13
  day 14 score 5: number analyzed (Participants) | 142 | 67
  day 14 score 5 | 17 | 10
  day 14 score 6: number analyzed (Participants) | 142 | 67
  day 14 score 6 | 4 | 4
  day 14 score 7: number analyzed (Participants) | 142 | 67
  day 14 score 7 | 2 | 1
  day 21 score 1: number analyzed (Participants) | 121 | 55
  day 21 score 1 | 74 | 36
  day 21 score 2: number analyzed (Participants) | 121 | 55
  day 21 score 2 | 8 | 2
  day 21 score 3: number analyzed (Participants) | 121 | 55
  day 21 score 3 | 13 | 5
  day 21 score 4: number analyzed (Participants) | 121 | 55
  day 21 score 4 | 14 | 5
  day 21 score 5: number analyzed (Participants) | 121 | 55
  day 21 score 5 | 6 | 5
  day 21 score 6: number analyzed (Participants) | 121 | 55
  day 21 score 6 | 5 | 0
  day 21 score 7: number analyzed (Participants) | 121 | 55
  day 21 score 7 | 1 | 2
  HD score 1: number analyzed (Participants) | 134 | 61
  HD score 1 | 11 | 6
  HD score 2: number analyzed (Participants) | 134 | 61
  HD score 2 | 2 | 4
  HD score 3: number analyzed (Participants) | 134 | 61
  HD score 3 | 109 | 48
  HD score 4: number analyzed (Participants) | 134 | 61
  HD score 4 | 10 | 3
  HD score 5: number analyzed (Participants) | 134 | 61
  HD score 5 | 0 | 0
  HD score 6: number analyzed (Participants) | 134 | 61
  HD score 6 | 0 | 0
  HD score 7: number analyzed (Participants) | 134 | 61
  HD score 7 | 0 | 0
  day 28 score 1: number analyzed (Participants) | 131 | 59
  day 28 score 1 | 100 | 40
  day 28 score 2: number analyzed (Participants) | 131 | 59
  day 28 score 2 | 8 | 8
  day 28 score 3: number analyzed (Participants) | 131 | 59
  day 28 score 3 | 7 | 1
  day 28 score 4: number analyzed (Participants) | 131 | 59
  day 28 score 4 | 8 | 5
  day 28 score 5: number analyzed (Participants) | 131 | 59
  day 28 score 5 | 2 | 2
  day 28 score 6: number analyzed (Participants) | 131 | 59
  day 28 score 6 | 4 | 2
  day 28 score 7: number analyzed (Participants) | 131 | 59
  day 28 score 7 | 2 | 1
  EoT score 1: number analyzed (Participants) | 164 | 77
  EoT score 1 | 3 | 2
  EoT score 2: number analyzed (Participants) | 164 | 77
  EoT score 2 | 0 | 0
  EoT score 3: number analyzed (Participants) | 164 | 77
  EoT score 3 | 92 | 36
  EoT score 4: number analyzed (Participants) | 164 | 77
  EoT score 4 | 36 | 18
  EoT score 5: number analyzed (Participants) | 164 | 77
  EoT score 5 | 25 | 15
  EoT score 6: number analyzed (Participants) | 164 | 77
  EoT score 6 | 7 | 5
  EoT score 7: number analyzed (Participants) | 164 | 77
  EoT score 7 | 1 | 1
  Day 60 score 1: number analyzed (Participants) | 136 | 65
  Day 60 score 1 | 125 | 56
  Day 60 score 2: number analyzed (Participants) | 136 | 65
  Day 60 score 2 | 9 | 6
  Day 60 score 3: number analyzed (Participants) | 136 | 65
  Day 60 score 3 | 1 | 0
  Day 60 score 4: number analyzed (Participants) | 136 | 65
  Day 60 score 4 | 0 | 1
  Day 60 score 5: number analyzed (Participants) | 136 | 65
  Day 60 score 5 | 1 | 2
  Day 60 score 6: number analyzed (Participants) | 136 | 65
  Day 60 score 6 | 0 | 0
  Day 60 score 7: number analyzed (Participants) | 136 | 65
  Day 60 score 7 | 0 | 0
  Day 90 score 1: number analyzed (Participants) | 14 | 4
  Day 90 score 1 | 14 | 4
  Day 90 score 2: number analyzed (Participants) | 14 | 4
  Day 90 score 2 | 0 | 0
  Day 90 score 3: number analyzed (Participants) | 14 | 4
  Day 90 score 3 | 0 | 0
  Day 90 score 4: number analyzed (Participants) | 14 | 4
  Day 90 score 4 | 0 | 0
  Day 90 score 5: number analyzed (Participants) | 14 | 4
  Day 90 score 5 | 0 | 0
  Day 90 score 6: number analyzed (Participants) | 14 | 4
  Day 90 score 6 | 0 | 0
  Day 90 score 7: number analyzed (Participants) | 14 | 4
  Day 90 score 7 | 0 | 0
  EoS score 1: number analyzed (Participants) | 154 | 75
  EoS score 1 | 132 | 57
  EoS score 2: number analyzed (Participants) | 154 | 75
  EoS score 2 | 7 | 6
  EoS score 3: number analyzed (Participants) | 154 | 75
  EoS score 3 | 1 | 0
  EoS score 4: number analyzed (Participants) | 154 | 75
  EoS score 4 | 2 | 1
  EoS score 5: number analyzed (Participants) | 154 | 75
  EoS score 5 | 3 | 4
  EoS score 6: number analyzed (Participants) | 154 | 75
  EoS score 6 | 1 | 2
  EoS score 7: number analyzed (Participants) | 154 | 75
  EoS score 7 | 8 | 5
Statistical Analysis 1: Comparison: Reparixin vs Placebo; day 3 - please note that the number of subjects in this analysis is not 270 but 255; Test type: Superiority; p = 0.444, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Reparixin vs Placebo; day 7 - please note that the number of subjects in this analysis is not 270 but 246; Test type: Superiority; p = 0.357, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Reparixin vs Placebo; day 14 - please note that the number of subjects in this analysis is not 270 but 209; Test type: Superiority; p = 0.484, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Reparixin vs Placebo; day 21 - please note that the number of subjects in this analysis is not 270 but 176; Test type: Superiority; p = 0.753, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Reparixin vs Placebo; day 28 - please note that the number of subjects in this analysis is not 270 but 190; Test type: Superiority; p = 0.26, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Reparixin vs Placebo; day 60 - please note that the number of subjects in this analysis is not 270 but 201; Test type: Superiority; p = 0.19, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Reparixin vs Placebo; day 90 - please note that the number of subjects in this analysis is not 270 but 18; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Reparixin vs Placebo; EOS - please note that the number of subjects in this analysis is not 270 but 229; Test type: Superiority; p = 0.074, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Reparixin vs Placebo; EOT - please note that the number of subjects in this analysis is not 270 but 241; Test type: Superiority; p = 0.193, two-sample Mann-Whitney U test
Statistical Analysis 10: Comparison: Reparixin vs Placebo; Hospital discharge - please note that the number of subjects in this analysis is not 270 but 195; Test type: Superiority; p = 0.131, two-sample Mann-Whitney U test

14. Secondary Outcome: The Number of Patients With Different Dyspnea Severity Scores Using the Likert Scale at Fixed Timepoints
Description: The number of patients with Dyspnea severity Likert scale by score and treatment group is calculated for each time point.
  Likert scale: grading the current experience of breathing discomfort compared to baseline (randomization) status (from -3 to 3) where:
  "-1 = minimally worse; -2 = moderately worse; -3 = markedly worse; 0 = no change; 1 = minimally better; 2 = moderately better; 3 = markedly better" More negative the score, the worse the outcome.
Time Frame: as for outcome 7
Population: FAS Full Analysis Set: set which consisted of all randomized subjects who received at least one dose of the IMP.
Measure: Number; unit: participants
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 182 | 88
participants
  day 3 score -3: number analyzed (Participants) | 103 | 52
  day 3 score -3 | 1 | 0
  day 3 score -2: number analyzed (Participants) | 103 | 52
  day 3 score -2 | 1 | 3
  day 3 score -1: number analyzed (Participants) | 103 | 52
  day 3 score -1 | 5 | 1
  day 3 score 0: number analyzed (Participants) | 103 | 52
  day 3 score 0 | 22 | 10
  day 3 score 1: number analyzed (Participants) | 103 | 52
  day 3 score 1 | 37 | 18
  day 3 score 2: number analyzed (Participants) | 103 | 52
  day 3 score 2 | 26 | 17
  day 3 score 3: number analyzed (Participants) | 103 | 52
  day 3 score 3 | 11 | 3
  day 7 score -3: number analyzed (Participants) | 96 | 47
  day 7 score -3 | 1 | 0
  day 7 score -2: number analyzed (Participants) | 96 | 47
  day 7 score -2 | 0 | 1
  day 7 score -1: number analyzed (Participants) | 96 | 47
  day 7 score -1 | 0 | 1
  day 7 score 0: number analyzed (Participants) | 96 | 47
  day 7 score 0 | 9 | 6
  day 7 score 1: number analyzed (Participants) | 96 | 47
  day 7 score 1 | 19 | 8
  day 7 score 2: number analyzed (Participants) | 96 | 47
  day 7 score 2 | 31 | 13
  day 7 score 3: number analyzed (Participants) | 96 | 47
  day 7 score 3 | 36 | 18
  day 14 score -3: number analyzed (Participants) | 76 | 39
  day 14 score -3 | 0 | 0
  day 14 score -2: number analyzed (Participants) | 76 | 39
  day 14 score -2 | 2 | 0
  day 14 score -1: number analyzed (Participants) | 76 | 39
  day 14 score -1 | 0 | 0
  day 14 score 0: number analyzed (Participants) | 76 | 39
  day 14 score 0 | 9 | 1
  day 14 score 1: number analyzed (Participants) | 76 | 39
  day 14 score 1 | 6 | 6
  day 14 score 2: number analyzed (Participants) | 76 | 39
  day 14 score 2 | 18 | 7
  day 14 score 3: number analyzed (Participants) | 76 | 39
  day 14 score 3 | 41 | 25
  day 21 score -3: number analyzed (Participants) | 60 | 32
  day 21 score -3 | 1 | 0
  day 21 score -2: number analyzed (Participants) | 60 | 32
  day 21 score -2 | 0 | 0
  day 21 score -1: number analyzed (Participants) | 60 | 32
  day 21 score -1 | 0 | 0
  day 21 score 0: number analyzed (Participants) | 60 | 32
  day 21 score 0 | 6 | 3
  day 21 score 1: number analyzed (Participants) | 60 | 32
  day 21 score 1 | 9 | 2
  day 21 score 2: number analyzed (Participants) | 60 | 32
  day 21 score 2 | 9 | 7
  day 21 score 3: number analyzed (Participants) | 60 | 32
  day 21 score 3 | 35 | 20
  HD score -3: number analyzed (Participants) | 38 | 27
  HD score -3 | 0 | 0
  HD score -2: number analyzed (Participants) | 38 | 27
  HD score -2 | 0 | 1
  HD score -1: number analyzed (Participants) | 38 | 27
  HD score -1 | 0 | 0
  HD score 0: number analyzed (Participants) | 38 | 27
  HD score 0 | 2 | 2
  HD score 1: number analyzed (Participants) | 38 | 27
  HD score 1 | 3 | 1
  HD score 2: number analyzed (Participants) | 38 | 27
  HD score 2 | 5 | 4
  HD score 3: number analyzed (Participants) | 38 | 27
  HD score 3 | 28 | 19
  day 28 score -3: number analyzed (Participants) | 73 | 33
  day 28 score -3 | 0 | 0
  day 28 score -2: number analyzed (Participants) | 73 | 33
  day 28 score -2 | 0 | 0
  day 28 score -1: number analyzed (Participants) | 73 | 33
  day 28 score -1 | 0 | 0
  day 28 score 0: number analyzed (Participants) | 73 | 33
  day 28 score 0 | 9 | 3
  day 28 score 1: number analyzed (Participants) | 73 | 33
  day 28 score 1 | 7 | 3
  day 28 score 2: number analyzed (Participants) | 73 | 33
  day 28 score 2 | 9 | 7
  day 28 score 3: number analyzed (Participants) | 73 | 33
  day 28 score 3 | 48 | 20
  EoT score -3: number analyzed (Participants) | 77 | 38
  EoT score -3 | 3 | 0
  EoT score -2: number analyzed (Participants) | 77 | 38
  EoT score -2 | 1 | 0
  EoT score -1: number analyzed (Participants) | 77 | 38
  EoT score -1 | 0 | 1
  EoT score 0: number analyzed (Participants) | 77 | 38
  EoT score 0 | 4 | 0
  EoT score 1: number analyzed (Participants) | 77 | 38
  EoT score 1 | 12 | 7
  EoT score 2: number analyzed (Participants) | 77 | 38
  EoT score 2 | 17 | 6
  EoT score 3: number analyzed (Participants) | 77 | 38
  EoT score 3 | 40 | 24
  EOS score -3: number analyzed (Participants) | 2 | 0
  EOS score -3 | 0 |
  EOS score -2: number analyzed (Participants) | 2 | 0
  EOS score -2 | 0 |
  EOS score -1: number analyzed (Participants) | 2 | 0
  EOS score -1 | 0 |
  EOS score 0: number analyzed (Participants) | 2 | 0
  EOS score 0 | 1 |
  EOS score 1: number analyzed (Participants) | 2 | 0
  EOS score 1 | 1 |
  EOS score 2: number analyzed (Participants) | 2 | 0
  EOS score 2 | 0 |
  EOS score 3: number analyzed (Participants) | 2 | 0
  EOS score 3 | 0 |
Statistical Analysis 1: Comparison: Reparixin vs Placebo; at day 3 - Please note that the number of subjects in this analysis is not 270 but 155; Test type: Superiority; p = 0.997, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Reparixin vs Placebo; at day 7 - Please note that the number of subjects in this analysis is not 270 but 143; Test type: Superiority; p = 0.712, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Reparixin vs Placebo; at day 14 - Please note that the number of subjects in this analysis is not 270 but 115; Test type: Superiority; p = 0.241, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Reparixin vs Placebo; at day 21 - Please note that the number of subjects in this analysis is not 270 but 92; Test type: Superiority; p = 0.528, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Reparixin vs Placebo; at day 28 - Please note that the number of subjects in this analysis is not 270 but 106; Test type: Superiority; p = 0.814, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Reparixin vs Placebo; at EOT - Please note that the number of subjects in this analysis is not 270 but 115; Test type: Superiority; p = 0.242, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Reparixin vs Placebo; at hospital discharge (HD) - Please note that the number of subjects in this analysis is not 270 but 65; Test type: Superiority; p = 0.722, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Change From Baseline to Fixed Timepoints in Pulse Oximetry by Measurement of Peripheral Arterial Oxygen Saturation (SpO2).
Description: Peripheral oxygen saturation (SpO2) monitoring by pulse oximetry is used to estimate the oxygen saturation of arterial blood (SaO2) and provides vital information about a patient's cardiorespiratory function.
Time Frame: as for outcome 7
Population: The Full Analysis Set (FAS), which consisted of all randomized subjects who received at least one dose of the IMP.
Measure: Mean (Standard Deviation); unit: percentage of oxygenated hemoglobin
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 182 | 88
percentage of oxygenated hemoglobin
  Day 3: number analyzed (Participants) | 166 | 80
  Day 3 | 0.79 (2.88) | 0.36 (2.78)
  Day 7: number analyzed (Participants) | 151 | 74
  Day 7 | 0.76 (2.89) | 0.49 (3.38)
  Day 14: number analyzed (Participants) | 75 | 43
  Day 14 | 0.46 (2.93) | -0.83 (3.99)
  Day 21: number analyzed (Participants) | 35 | 19
  Day 21 | -0.85 (4.92) | -5.35 (11.82)
  Day 28: number analyzed (Participants) | 22 | 10
  Day 28 | -0.99 (6.15) | -1.56 (6.78)
  day 60 EoS: number analyzed (Participants) | 1 | 2
  day 60 EoS | -2.70 (000) | -2.00 (0.00)
  EoT: number analyzed (Participants) | 145 | 67
  EoT | 0.24 (2.69) | -0.68 (3.76)
  HD: number analyzed (Participants) | 102 | 50
  HD | 0.57 (2.60) | 0.28 (2.76)
  EoS: number analyzed (Participants) | 7 | 7
  EoS | -7.57 (11.12) | -11.01 (18.49)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; at day 3 - Please note that the number of subjects in this analysis is not 270, but it is 246; Test type: Superiority; p = 0.053, two-sample Mann-Whitney U test
Statistical Analysis 2: Comparison: Reparixin vs Placebo; at day 7 - Please note that the number of subjects in this analysis is not 270, but it is 225; Test type: Superiority; p = 0.245, two-sample Mann-Whitney U test
Statistical Analysis 3: Comparison: Reparixin vs Placebo; at day 14 - Please note that the number of subjects in this analysis is not 270, but it is 118; Test type: Superiority; p = 0.067, two-sample Mann-Whitney U test
Statistical Analysis 4: Comparison: Reparixin vs Placebo; at day 21 - Please note that the number of subjects in this analysis is not 270, but it is 54; Test type: Superiority; p = 0.051, two-sample Mann-Whitney U test
Statistical Analysis 5: Comparison: Reparixin vs Placebo; at day 28 - Please note that the number of subjects in this analysis is not 270, but it is 32; Test type: Superiority; p = 0.684, two-sample Mann-Whitney U test
Statistical Analysis 6: Comparison: Reparixin vs Placebo; at EOS - Please note that the number of subjects in this analysis is not 246, but it is 14; Test type: Superiority; p = 1.00, two-sample Mann-Whitney U test
Statistical Analysis 7: Comparison: Reparixin vs Placebo; at Day 60 - Please note that the number of subjects in this analysis is not 246, but it is 3; Test type: Superiority; p = 0.48, two-sample Mann-Whitney U test
Statistical Analysis 8: Comparison: Reparixin vs Placebo; at Hospital discharge - Please note that the number of subjects in this analysis is 152; Test type: Superiority; p = 0.638, two-sample Mann-W hitney U test
Statistical Analysis 9: Comparison: Reparixin vs Placebo; at EoT - Please note that the number of subjects in this analysis is 212; Test type: Superiority; p = 0.137, two-sample Mann-W hitney U test

16. Secondary Outcome: Change From Baseline in Dyspnea Severity (VAS Scale) at Fixed Timepoints
Description: The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between paints with similar conditions.The VAS scale is from 0 to 100. The number 0 means the worst breathing the patient has ever felt, and the number 100 means the best the patient has ever felt.
Time Frame: as for outcome 7
Population: FAS Full Analysis Set: set which consisted of all randomized subjects who received at least one dose of the IMP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 182 | 88
score on a scale
  day 3: number analyzed (Participants) | 105 | 52
  day 3 | 6.4 (25.3) | 2.2 (20.6)
  day 7 (+/-1): number analyzed (Participants) | 93 | 46
  day 7 (+/-1) | 8.3 (31.1) | -0.2 (31.1)
  day 14(+/-2): number analyzed (Participants) | 46 | 27
  day 14(+/-2) | 12.7 (38.5) | 6.6 (37.4)
  day 21 (+/-2): number analyzed (Participants) | 15 | 8
  day 21 (+/-2) | 16.0 (39.5) | 32.5 (14.3)
  day 28 (+/-2): number analyzed (Participants) | 14 | 3
  day 28 (+/-2) | 31.1 (20.3) | 40.7 (8.3)
  Hospital discharge: number analyzed (Participants) | 38 | 20
  Hospital discharge | 12.3 (44.0) | 10.2 (41.5)
  EoT: number analyzed (Participants) | 77 | 36
  EoT | 17.1 (32.6) | 8.6 (37.8)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; at day 3 - Please note that the number of subjects in this analysis is not 270, but it is 157; Test type: Superiority; p = 0.399, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Reparixin vs Placebo; at day 7 - Please note that the number of subjects in this analysis is not 270, but it is 139; Test type: Superiority; p = 0.07, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Reparixin vs Placebo; at day 14 - Please note that the number of subjects in this analysis is not 270, but it is 73; Test type: Superiority; p = 0.4, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Reparixin vs Placebo; at day 21 - Please note that the number of subjects in this analysis is not 270, but it is 23; Test type: Superiority; p = 0.517, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Reparixin vs Placebo; at day 28 - Please note that the number of subjects in this analysis is not 270, but it is 17; Test type: Superiority; p = 0.445, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Reparixin vs Placebo; at EoT - Please note that the number of subjects in this analysis is not 270, but it is 113; Test type: Superiority; p = 0.324, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Reparixin vs Placebo; at Hospital discharge - Please note that the number of subjects in this analysis is not 270, but it is 67; Test type: Superiority; p = 0.752, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Duration of Supplemental Oxygen Treatment up to Day 28
Description: This endpoint is expressed as:
  * The number and proportion along with the 95% CI (Clopper-Pearson's formula) of patients using supplemental oxygen treatment by treatment group;
  * The Cumulative duration of supplemental oxygen treatment in days analyzed by means of descriptive statistics by treatment. This latter is reported in the system.
Time Frame: From baseline up to day 28
Population: FAS population is used in this table. Discrepancies between the total number of patients in the FAS and patients actually analyzed in the model are due to the presence of missing data for which no imputation methods are expected for this endpoint.
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 174 | 81
day | 10.5 (7.3) | 10.8 (6.8)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Please note that the number of patients in this analysis is not 270 but 255, because patients who used supplement oxygen were 174 in the Reparixin group and 81 in the placebo group; Test type: Superiority; p = 0.447, two-sample Mann-Whitney U test

18. Secondary Outcome: Number of Patients Requiring Invasive Mechanical Ventilation Use, or ECMO up to Day 28 and up to Day 60
Description: Invasive mechanical ventilation is defined as the delivery of positive pressure to the lungs via an endotracheal or tracheostomy tube. During mechanical ventilation, a predetermined mixture of air (ie, oxygen and other gases) is forced into the central airways and then flows into the alveoli.
Time Frame: day 28 and Day 60
Population: FAS population is used in this table. Discrepancies between the total number of patients in the FAS and patients actually analyzed in the model at Day 28 are due to the presence of missing data for which no imputation methods are expected for this endpoint.
Measure: Number; unit: Number of patient with event
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 182 | 88
Number of patient with event
  Up to day 28: number analyzed (Participants) | 163 | 82
  Up to day 28 | 9 | 10
  Up to day 60 | 9 | 10
Statistical Analysis 1: Comparison: Reparixin vs Placebo; At day 28 - Please note that the number of patients in this analysis is not 270 but 245, because patients requiring IMV or ECMO were 163 in the Reparixin group and 82 in the placebo group; Test type: Superiority; p = 0.065, Chi-squared — Comparison between treatment arms is performed by means of a Chi-squared test
Statistical Analysis 2: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.072, Chi-squared; Comparison between treatment arms is performed by means of a Chi-squared test

19. Secondary Outcome: Duration of Non-invasive Mechanical Ventilation up to Day 60
Description: Non-invasive ventilation (NIV) is the delivery of oxygen (ventilation support) via a face mask and therefore eliminating the need of an endotracheal airway. NIV achieves comparative physiological benefits to conventional mechanical ventilation by reducing the work of breathing and improving gas exchange.
Time Frame: From baseline up to day 60
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 66 | 32
days | 9.0 (7.9) | 10.1 (7.5)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.485, two-sample Mann-Whitney U test — Number of subjects included in analysis: 98

20. Secondary Outcome: Duration of Invasive Mechanical Ventilation, or ECMO up to Day 60
Description: as for outcome 18
Time Frame: Up to day 60
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 9 | 9
Days | 24.8 (16.8) | 15.9 (13.9)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Number of subjects included in analysis: 17; Test type: Superiority; p = 0.267, two-sample Mann-Whitney U test

21. Secondary Outcome: Duration of ICU Admission up to Day 60
Description: Admission to intensive care unit or ICU is linked to worsening of respiratory parameters compared to baseline.
Time Frame: Up to day 60
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 12 | 12
Days | 17.9 (10.1) | 11.4 (6.7)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority; p = 0.137, two-sample Mann-Whitney U test

22. Secondary Outcome: Change From Baseline to Fixed Timepoints of Partial Pressure of Oxygen (PaO2)
Description: PaO2-the oxygen pressure in arterial blood. The PaO2 reflects how well oxygen is able to move from the lungs to the blood. It is often altered by severe illnesses, with the PaO2 test results used to guide treatment.
Time Frame: as for outcome 7
Population: The Full Analysis Set (FAS), which consisted of all randomized subjects who received at least one dose of the IMP.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 182 | 88
mmHg
  Day 3: number analyzed (Participants) | 111 | 57
  Day 3 | 13.377 (36.568) | -5.274 (41.103)
  Day 7: number analyzed (Participants) | 99 | 47
  Day 7 | 3.147 (33.541) | 12.777 (81.367)
  Day 14: number analyzed (Participants) | 48 | 28
  Day 14 | 4.002 (54.235) | -7.257 (50.645)
  Day 21: number analyzed (Participants) | 24 | 14
  Day 21 | 3.388 (43.520) | -14.014 (54.603)
  Day 28: number analyzed (Participants) | 16 | 7
  Day 28 | -6.700 (31.896) | -52.171 (76.278)
  HD: number analyzed (Participants) | 48 | 26
  HD | -3.633 (29.723) | -8.869 (37.953)
  EOT: number analyzed (Participants) | 87 | 44
  EOT | 3.020 (50.296) | -7.189 (55.550)
  EOS: number analyzed (Participants) | 4 | 4
  EOS | 1.825 (20.570) | 51.950 (215.446)
  Day 60: number analyzed (Participants) | 1 | 0
  Day 60 | 1 (73.000) |
Statistical Analysis 1: Comparison: Reparixin vs Placebo; at day 3 - Please note that the number of subjects in this analysis is 168; Test type: Superiority; p = 0.002, two-sample Mann-Whitney U test
Statistical Analysis 2: Comparison: Reparixin vs Placebo; at day 7 - Please note that the number of subjects in this analysis is not 168, but it is 146; Test type: Superiority; p = 0.943, two-sample Mann-Whitney U test
Statistical Analysis 3: Comparison: Reparixin vs Placebo; at day 14 - Please note that the number of subjects in this analysis is not 168, but it is 76; Test type: Superiority; p = 0.88, two-sample Mann-Whitney U test
Statistical Analysis 4: Comparison: Reparixin vs Placebo; at day 21 - Please note that the number of subjects in this analysis is not 168, but it is 38; Test type: Superiority; p = 0.458, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Reparixin vs Placebo; at day 28 - Please note that the number of subjects in this analysis is not 168, but it is 23; Test type: Superiority; p = 0.285, two-sample Mann-Whitney U test
Statistical Analysis 6: Comparison: Reparixin vs Placebo; at EOS - Please note that the number of subjects in this analysis is not 168, but it is 8; Test type: Superiority; p = 0.885, two-sample Mann-Whitney U test
Statistical Analysis 7: Comparison: Reparixin vs Placebo; at HD - Please note that the number of subjects in this analysis is not 270, but it is 74; Test type: Superiority; p = 0.583, two-sample Mann-Whitney U test
Statistical Analysis 8: Comparison: Reparixin vs Placebo; at End of treatment - Please note that the number of subjects in this analysis is not 270, but it is 131; Test type: Superiority; p = 0.5, two-sample Mann-Whitney U test

23. Secondary Outcome: Change From Baseline to Fixed Timepoints in PaO2/FiO2 Ratio.
Description: The PaO2/FiO2 ratio is used to determine the severity of lung injury in mechanically ventilated patients.
  A normal P/F Ratio is ≥ 400 and equivalent to a PaO2 ≥ 80 mmHg on room air. Low values of the PaO2/FIO2 ratio may be due to pathological conditions, primarily those of a respiratory nature (atelectasis, ARDS, acute pulmonary edema, pneumonia, etc.), as well as to alterations in hemodynamic status (cardiogenic shock, septic shock, etc.), or even both.
Time Frame: as for outcome 7
Population: The Full Analysis Set (FAS), which consisted of all randomized subjects who received at least one dose of the IMP.
Measure: Mean (Standard Deviation); unit: PaO2/FiO2 Ratio
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 182 | 88
PaO2/FiO2 Ratio
  Day 3: number analyzed (Participants) | 163 | 82
  Day 3 | 30.329 (81.291) | 0.398 (87.607)
  Day 7 ± 1: number analyzed (Participants) | 148 | 73
  Day 7 ± 1 | 77.528 (106.383) | 65.291 (138.832)
  Day 14 ± 2: number analyzed (Participants) | 74 | 43
  Day 14 ± 2 | 127.111 (135.063) | 111.220 (171.013)
  Day 21 ± 2: number analyzed (Participants) | 31 | 20
  Day 21 ± 2 | 122.746 (114.603) | 62.520 (163.712)
  EoT: number analyzed (Participants) | 140 | 66
  EoT | 140.575 (139.619) | 106.332 (144.608)
  Day 28 ± 2: number analyzed (Participants) | 21 | 8
  Day 28 ± 2 | 145.043 (146.515) | -22.125 (123.435)
  HD (hospital discharge): number analyzed (Participants) | 96 | 48
  HD (hospital discharge) | 228.999 (119.337) | 210.765 (112.418)
  Day 60 ± 2: number analyzed (Participants) | 1 | 2
  Day 60 ± 2 | 200.000 (000) | 334.000 (53.740)
  EOS: number analyzed (Participants) | 6 | 7
  EOS | -5.333 (89.844) | -30.714 (191.669)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; at day 3 - Please note that the number of subjects in this analysis is not 270, but it is 245; Test type: Superiority; p = 0.005, Mann-Whitney U test — Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test
Statistical Analysis 2: Comparison: Reparixin vs Placebo; at day 7 - Please note that the number of subjects in this analysis is not 270, but it is 221; Test type: Superiority; p = 0.283, Mann-Whitney U test — Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test
Statistical Analysis 3: Comparison: Reparixin vs Placebo; at day 14 - Please note that the number of subjects in this analysis is not 270, but it is 117; Test type: Superiority; p = 0.512, Mann-Whitney U test — Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test
Statistical Analysis 4: Comparison: Reparixin vs Placebo; at day 21 - Please note that the number of subjects in this analysis is not 270, but it is 51; Test type: Superiority; p = 0.174, Mann-Whitney U test; Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test
Statistical Analysis 5: Comparison: Reparixin vs Placebo; Test type: Superiority — at EOT - Please note that the number of subjects in this analysis is not 270, but it is 206; p = 0.133, Mann-Whitney U test; Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test
Statistical Analysis 6: Comparison: Reparixin vs Placebo; at day 28 ± 2 - Please note that the number of subjects in this analysis is not 270, but it is 29; Test type: Superiority; p = 0.009, Mann-Whitney U test; Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test
Statistical Analysis 7: Comparison: Reparixin vs Placebo; to HD - Please note that the number of subjects in this analysis is not 270, but it is 144; Test type: Superiority; p = 0.593, Mann-Whitney U test; Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test
Statistical Analysis 8: Comparison: Reparixin vs Placebo; to day 60 - Please note that the number of subjects in this analysis is not 270, but it is 3; Test type: Superiority; p = 0.540, Mann-Whitney U test; Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test
Statistical Analysis 9: Comparison: Reparixin vs Placebo; to EOS - Please note that the number of subjects in this analysis is not 270, but it is 13; Test type: Superiority; p = 0.224, Mann-Whitney U test; Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test

24. Secondary Outcome: Change From Baseline to Fixed Endpoints in High-Sensitivity C Reactive Protein (Hs-CRP)
Description: The high-sensitivity C-reactive protein (hs-CRP) test is more sensitive than the standard CRP test measuring slight increases in CRP levels even when within the normal range. Because of this greater sensitivity, the hs-CRP test can help determine your risk of cardiovascular disease (CVD).
Time Frame: as for outcome 7
Population: FAS population is used in this table. Discrepancies between the total number of patients in the FAS and patients actually analyzed in the model are due to the presence of missing data for which no imputation methods are expected for this endpoint. Please note that the Number Analyzed per Row includes those participants who contributed data at the specified time point.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 46 | 31
mg/L
  Day 3: number analyzed (Participants) | 9 | 6
  Day 3 | -30.7 (23.13) | -21.67 (53.33)
  Day 7 ± 1: number analyzed (Participants) | 8 | 5
  Day 7 ± 1 | -25.90 (95.74) | -29.62 (37.85)
  Day 14 ± 2: number analyzed (Participants) | 8 | 5
  Day 14 ± 2 | -25.21 (66.53) | -45.24 (62.83)
  Day 21 ± 2: number analyzed (Participants) | 5 | 4
  Day 21 ± 2 | -27.50 (72.23) | -47.05 (99.48)
  EOT: number analyzed (Participants) | 7 | 6
  EOT | 37.50 (151.54) | -37.68 (76.26)
  Day 28 ± 2: number analyzed (Participants) | 4 | 2
  Day 28 ± 2 | -42.60 (30.15) | 9.65 (26.94)
  HD (hospital discharge): number analyzed (Participants) | 5 | 3
  HD (hospital discharge) | -54.46 (63.12) | -84.83 (76.02)
Statistical Analysis 1: Comparison: Reparixin vs Placebo; to day 3 - Please note that the number of subjects in this analysis is not 270, but it is 15; Test type: Superiority; p = 0.68, Mann-Whitney U test; Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test
Statistical Analysis 2: Comparison: Reparixin vs Placebo; to day 7 - Please note that the number of subjects in this analysis is not 270, but it is 13; Test type: Superiority; p = 0.272, Mann-Whitney U test — Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test
Statistical Analysis 3: Comparison: Reparixin vs Placebo; to day 14 - Please note that the number of subjects in this analysis is not 270, but it is 13; Test type: Superiority; p = 1.000, Mann-Whitney U test — Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test
Statistical Analysis 4: Comparison: Reparixin vs Placebo; to day 21 - Please note that the number of subjects in this analysis is not 270, but it is 9; Test type: Superiority; p = 0.903, Mann-Whitney U test — Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test
Statistical Analysis 5: Comparison: Reparixin vs Placebo; to EOT - Please note that the number of subjects in this analysis is not 270, but it is 13; Test type: Superiority; p = 0.432, Mann-Whitney U test — Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test
Statistical Analysis 6: Comparison: Reparixin vs Placebo; to day 28 - Please note that the number of subjects in this analysis is not 270, but it is 6; Test type: Superiority; p = 0.105, Mann-Whitney U test — Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test
Statistical Analysis 7: Comparison: Reparixin vs Placebo; to HD - Please note that the number of subjects in this analysis is not 270, but it is 8; Test type: Superiority; p = 0.551, Mann-Whitney U test — Comparison between treatment arms is performed by means of two-sample Mann-Whitney U test

25. Secondary Outcome: Mortality Rates up to Days 60 and 90
Description: Mortality rate, or death rate, is a measure of the number of deaths (in general, or due to a specific cause) in a particular population, scaled to the size of that population, per unit of time. The death event variable is defined as the proportion of patients died up to Day 90.
Time Frame: up to Days 60 and 90
Population: as for outcome 17
Measure: Number; unit: dead patients
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 182 | 88
dead patients
  Day 60: number analyzed (Participants) | 156 | 76
  Day 60 | 11 | 7
  Day 90: number analyzed (Participants) | 27 | 12
  Day 90 | 11 | 7
Statistical Analysis 1: Comparison: Reparixin vs Placebo; up to day 60; Test type: Superiority; p = 0.232, Regression, Logistic — Analysis is based on logistic regression model with proportion of patients died up to Day 60 as dependent variable, treatment, age group, gender and presence of concomitant disease at baseline as qualitative independent variables; Odds Ratio (OR) = 0.520, 95% CI 2-sided [0.178 to 1.522]
Statistical Analysis 2: Comparison: Reparixin vs Placebo; Up to Day 90; Test type: Superiority — Analysis is based on logistic regression model with proportion of patients died up to Day 90 as dependent variable, treatment, age group, gender and presence of concomitant disease at baseline as qualitative independent variables; p = 0.158, Regression, Logistic; Odds Ratio (OR) = 0.246, 95% CI 2-sided [0.034 to 1.782]

26. Secondary Outcome: Freedom From (Time to) Death or Respiratory Failure up to Day 90
Description: Freedom from (time to) death or respiratory failure (need of invasive mechanical ventilation or ECMO or admission to ICU linked to worsening of respiratory parameters compared to baseline) at baseline, day 3, day 7, day 14, day 21, day 28, day 60, day 90 was performed using the same Kaplan-Meier analysis and the one-sided log-rank test that were used to test for differences between groups.
Time Frame: at baseline, day 3, day 7, day 14, day 21, day 28, day 60, day 90
Population: The Full Analysis Set (FAS), which consisted of all randomized subjects who received at least one dose of the IMP.
Measure: Number; unit: participants with event
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 182 | 88
participants with event
  day 1 | 0 | 0
  day 3 | 2 | 1
  day 7 | 4 | 2
  day 14 | 9 | 5
  day 21 | 11 | 5
  day 28 | 16 | 6
  day 60 | 103 | 49
  day 90 | 154 | 72
Statistical Analysis 1: Comparison: Reparixin vs Placebo; Test type: Superiority — Freedom from (time to) death or respiratory failure (need of invasive mechanical ventilation or ECMO or admission to ICU linked to worsening of respiratory parameters compared to baseline) up to Day 90 was performed using the same Kaplan-Meier analysis and the one-sided log-rank test that were used to test for differences between groups; p = 0.33607, Log Rank

27. Secondary Outcome: Number of Subjects Who Exhibited at Least 1 TEAE, at Least 1 Severe TEAE, at Least 1 Serious TEAE, at Least 1 Non-serious TEAE, at Least 1 ADR, at Least 1 Serious ADR, at Least 1 TEAE Leading to Discontinuation of IMP, Etc.
Description: AE= An adverse event is any untoward or unfavorable medical occurrence in a human. subject, including any abnormal sign (for example, abnormal physical exam or. laboratory finding), symptom, or disease, temporally associated with the subject's.
  serious AE=a SAE iA serious adverse event (SAE) in human drug trials is defined as any untoward medical occurrence that at any dose results in death Is life-threatening Requires inpatient hospitalization or causes prolongation of existing hospitalization Results in persistent or significant disability/incapacity May have caused a congenital anomaly/birth defect Requires intervention to prevent permanent impairment or damage. The term "life-threatening" in the definition of "serious" refers to an event in which the patient was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe.
  Do note that starting from this point the safety endpoint is analysed.
Time Frame: Throughout the study, till Day 90 (= end of the follow-up period).
Population: The Safety set (SAF) consisted of all randomized subjects who received at least one dose of the IMP. The SAF population was analyzed according to the actual treatment received and was used to present results on safety data.
Measure: Number; unit: number of subjects
Arm/Group | Reparixin | Placebo
Number analyzed (Participants) | 182 | 88
number of subjects
  Number of Subjects with at least one TEAE | 83 | 48
  Number of Subjects with at least one serious TEAE | 20 | 13
  Number of Subjects with at least one severe TEAE | 16 | 12
  N. sub with at least 1TEAE leading to quit IMP | 19 | 11
  Number of subjects with at least 1TEAE leading to quit the study | 1 | 0
  Number of Subjects with TEAEs leading to death | 10 | 7

ADVERSE EVENTS:
Time Frame: From Baseline up to day 90 of the trial (=the end of the follow-up period).
Description: In the system AEs are reported for the overall period.
Groups:
- Reparixin SAF: Reparixin oral tablets, 1200 mg three times daily (TID) (2 tablets 600 mg each, TID) for up to 21 days or until decision of discharge from the hospital, on top of standard supportive care
  Reparixin: 2 tablets of Reparixin (600 mg each), for the total of three daily administrations (6 tablets daily).
  Please note that patients randomized to Reparixin were 185, but the ones receiving at least one dose of IMP were 182. Three patients, hence, in this group were excluded from the primary FAS analysis of efficacy and from the safety analysis.
- Placebo SAF: Placebo, 2 tablets TID (identical to Reparixin tablets) for up to 21 days or until decision of discharge from the hospital, on top of standard supportive care.
  For each administration, two tablets of Reparixin (600 mg each) or placebo were taken, for the total of three daily administrations (6 tablets daily). It was advisable to take the tablets with a glass of water to facilitate swallowing.
  Please note that patients randomized to placebo were 94, but the ones receiving it were 88. Six patients in this group, hence, were excluded from the primary FAS analysis of efficacy and from the safety analysis.
Arm/Group | Reparixin SAF | Placebo SAF
All-Cause Mortality (participants affected / at risk) | 11/182 | 7/88
Serious Adverse Events (participants affected / at risk) | 20/182 | 13/88
Other Adverse Events (participants affected / at risk) | 75/182 | 42/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reparixin SAF (N=182) | Placebo SAF (N=88)
Circulatory collapse (Vascular disorders) | 1 | 1
Thrombosis (Vascular disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 | 7
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Sepsis (Infections and infestations) | 2 | 1
Clostridium difficile infection (Infections and infestations) | 2 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reparixin SAF (N=182) | Placebo SAF (N=88)
Hypertension (Vascular disorders) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Poor venous access (Vascular disorders) | 1 (1) | 1 (1)
Thrombophlebitis (Vascular disorders) | 2 (2) | 0 (0)
Tracheostomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Illness (General disorders) | 3 (4) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 3 (4)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1)
Extravasation (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (7) | 4 (4)
Anxiety (Psychiatric disorders) | 5 (5) | 4 (4)
Agitation (Psychiatric disorders) | 3 (3) | 1 (1)
Mood altered (Psychiatric disorders) | 3 (5) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Persistent depressive disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Transaminases increased (Investigations) | 2 (2) | 1 (1)
Blood culture positive (Investigations) | 2 (2) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Culture urine positive (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Vitamin D decreased (Investigations) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 4 (5) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 1 (1)
Bradycadia (Cardiac disorders) | 3 (3) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (5) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Tinnitus (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 13 (14) | 10 (10)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 3 (3) | 2 (2)
Oliguria (Renal and urinary disorders) | 3 (3) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hyperparathyroidism secondary (Endocrine disorders) | 2 (2) | 0 (0)
Euthyroid sick syndrome (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Eating disorders (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Steroid diabetes (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 6 (6)
Pneumonia bacterial (Infections and infestations) | 4 (4) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 4 (4)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 2 (2)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Lower respiratory tract infection fungal (Infections and infestations) | 1 (1) | 1 (1)
Acquired immunodeficiency syndrome (Infections and infestations) | 0 (0) | 1 (1)
Anal infection (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Candida Infections (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus syndrome (Infections and infestations) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Moraxella infection (Infections and infestations) | 1 (1) | 0 (0)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Phlebitis infective (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT04878055/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/55/NCT04878055/SAP_002.pdf